CLINICAL TRIAL: NCT04006197
Title: Vocal Folds Irregular Mucosal Changes: A Clinical, Pathological and Genetic Study
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira Hafez Abdelaal, principal investigator, Assiut University
Other Study IDs: Vocal folds irregular mucosa
Record Dates: First submitted 2019-06-30; First posted 2019-07-05 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Vocal Cord Neoplasm
Keywords: vocal folds dysplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: laryngostroboscopy and histoh-pathology — videolaryngoscopy and laryngostroboscoby will be performed .the latter will be pathological in case of highly reduced or abolished amplitudes of vocal fold vibration and if there is reduction of mucosal wave propagation.also direct microlaryngoscopy under general anathesia will be done and excesional biobsy will be taken followed by histopatholpgical examination .the histological finding will be catagorized into the following categories according to (WHO): squamous cell hyperplasia with non dysplasia,mild dysplasia,moderate dysplasia,sever dysplasia,carcinoma in situ and squamous cell carcinoma.
  Other Names: 1.Telescopic orolaryngoscopic: 90○ rigid telescope R wolf (445057) - storz / Hopkins, 2.Tele pack X LED TP 100 storz.c)

SUMMARY:
simple combination of functional investigation, in form of laryngostroboscopy, together with conventional histopathological examination, provides a highly sensitive method in differential diagnosis of undiagnosed vocal folds irregularites

DETAILED DESCRIPTION:
Vocal folds irregular mucosal changes often manifest as mucosal surface changes of leukoplakia, erythroplakia and keratosis associated with tissue irregularities. Lesions that go beyond the outermost layer of the vocal fold and invade the intermediate and deep layers. These gross mucosal changes may represent benign, premalignant, or malignant entities as they correspond to large spectrum of lesions ranging from simple totally benign keratosis with or without atypia up to invasive carcinoma, it is commonly encountered in phoniatrics clinic and presents diagnostic and therapeutic challenge as there is no unified surgical indication or guidelines.

Laryngostroboscopy is very important and primary tool for assessment of morphological features and vibratory functions of the vocal folds. Stroboscopic evaluation allows early detection of infiltrative processes of the vocal folds. However, the laryngoscope examination may not always be sufficient to assess premalignant lesions and their exact delineation.

Gugatschka et al., 2008 reported that videostroboscopic evaluation allows early detection of infiltrative processes of the vocal folds, as they achieved a sensitivity of more than 97 %, when used a combination of cytology and videostroboscopy, in contrast to 74 % as found by cytology alone.

Zhang et al., 2018 proposed to classify VF leukoplakia into three types according to the morphological appearance. The evaluated features included texture, color, and thickness. They proved that type III-bulge and rough-with irregular, nonhomogeneous leukoplakia higher than mucosa surface was more often associated with cancerization or severe dysplasia in 29.3% and 21.5% cases, respectively, comparing to the respective percentages of 4.0% and 3.7% for type I-flat and smooth leukoplakia. Anna Rzepakowska et al submitted a protocol for evaluation of the morphological characteristics of leukoplakia which involved the following features of the lesion: color, texture, size, thickness, symmetry and vibratory function. Each character was assigned with the score of zero or one (score zero was considered to be a clinical indicator of benign lesions, while, score one was a clinical indicator of malignancy).

Recent advances in basic research have improved understanding of underlying mechanisms of molecular processes in early stages of laryngeal cancer development. The SOX2 gene located at 3q26 is frequently amplified and overexpressed in multiple cancers, including head and neck squamous cell carcinomas (HNSCC). The tumor-promoting activity and involvement of SOX2 in tumor progression has been extensively demonstrated, thereby emerging as a promising therapeutic target. However, the role of SOX2 in early stages of tumorigenesis and its possible contribution to malignant transformation remain unexplored. Granda-Diaz etal., 2019 investigated for the first time SOX2 gene in precancerous lesion using real-time PCR and demonstrated that SOX2 protein expression and gene amplification are frequent events in early stages of laryngeal tumorigenesis

ELIGIBILITY:
inclusion criteria

1. Age 18-70 years old males
2. Unilateral or bilateral localized and diffuse vocal fold irregularities.
3. Patients with white (leukoplakia) patches on one or both vocal folds
4. No previous microphonosurgery.
5. No previous history of radiotherapy .6.No impairment of the vocal fold mobility.

exclusion criteria

1. Subject refusal.
2. Patients with large exophytic and/or ulcerated mass.
3. Vocal fold cysts or polyps, contact granulomas, or Reinke's edema
4. If there is a concern for rapid growth pattern, airway obstruction requiring urgent operative intervention
5. Vocal fold immobility
6. History of allergies and GERD.
7. Unfit for general anesthesia

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: one hundred patient with localized or diffuse vocal folds irregularites wiii be examined for primary diagnosis at the phoniatric unit of ENT department in Assiut university hospital.main symptom of all patients is dysphonia of varying degree and dauration from afew days to several months .
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Correlation between video-stroboscopic examination and histopathological results | baseline
  Correlation between video-stroboscopic examination and histopathological groups.

SECONDARY OUTCOMES:
to correlate between SOX2 gene expression and histopathological finding | baseline
  to correlate between SOX2 gene expression and histopathological finding and if can give the same diagnosis of histopathology or not

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, faculty of medicine, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ferlito A, Devaney KO, Woolgar JA, Slootweg PJ, Paleri V, Takes RP, Strojan P, Bradley PJ, Rinaldo A. Squamous epithelial changes of the larynx: diagnosis and therapy. Head Neck. 2012 Dec;34(12):1810-6. doi: 10.1002/hed.21862. Epub 2011 Oct 3. PMID 21971762
- [Background] Gugatschka M, Kiesler K, Beham A, Rechenmacher J, Friedrich G. Hyperplastic epithelial lesions of the vocal folds: combined use of exfoliative cytology and laryngostroboscopy in differential diagnosis. Eur Arch Otorhinolaryngol. 2008 Jul;265(7):797-801. doi: 10.1007/s00405-007-0549-9. Epub 2007 Dec 4. PMID 18057948
- [Background] Sadri M, McMahon J, Parker A. Management of laryngeal dysplasia: a review. Eur Arch Otorhinolaryngol. 2006 Sep;263(9):843-52. doi: 10.1007/s00405-006-0078-y. Epub 2006 Jul 6. PMID 16823559